CLINICAL TRIAL: NCT05659238
Title: Impact of Exposure to Television and Electronic Devices on Attention and Language in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ann Gamal Yousef, Principle investigator, Assiut University
Other Study IDs: language development and TV
Record Dates: First submitted 2022-09-19; First posted 2022-12-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Language Development
Keywords: exposure to TV & electronics on language development

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: those who exposed early to TV (before 1 year age)with long time of exposure/day (6hours\day or more)
  Interventions: Behavioral: the effect on language development & attention
- 2: those who exposed later to TV (after 2 years of age) with short time of exposure/day.(2 hours \day or less)
  Interventions: Behavioral: the effect on language development & attention

INTERVENTIONS:
Behavioral: the effect on language development & attention — Tv & other electronic devices effects onn children's language development & attention

SUMMARY:
The objective is to examine association between TV exposure ,mobile device use and other electronic devices on attention and language development in children.

DETAILED DESCRIPTION:
During the last few years, the time spent in front of various screens including:TV Sets, vedio games, smart phones &computers has dramatically increased Television remains the predominant type of screen based activity among children.

Some studies showed that this trend has astrong negative influence on language development of children.

On the other hand.,other studies showed that infant directed informal computer use can be beneficial for language development in children.

Some studies proved that language development and vocabulary growth in young children are directly related to the amount of time parents spend speaking to them & also reported that on examining language perception learning &language production learning human human interactions had a strong influence on child's language development.

In spite of that, some parents believe that media content is educative for their children as increase their knowledge, other parents admitted to limiting their children's screen time to avoid conflict & social isolation or distract children as they encourage parent children education to reinforce their relationship with their children.

Other researches proved that young children who spend more time on touch screen devices were more likely to have emotional problems .

In this study the investigators will discuss the positive and negative effects of screen exposure on attention and langage development of children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged from 2-6 years collected from clinics of phoniatrics.
2. A questionnaire will be given to their mothers inquiring about

   1. the age of child at first exposure to TV or electronic devices .
   2. the time of exposure to TV or electronic devices /day
   3. duration of viewing TV or electronic devices from first exposure until participation of this study.

Exclusion Criteria:

1. IQ test less than 80 (any mental disabilities )
2. Hearing impairement .
3. physical or motor.
4. history of active language intervention before study.

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: So, the child will be classified into 2 groups :
  * group 1:those who exposed early to TV (before age of 1 year) with long time of exposure/day (6 hours/day) or more.
  * group 2:those who exposed later to TV (after age 2 years) with short time of exposure/day.(2 hours/day)or less.
  * Children in both groups will be matched in age ,sex, social status , & educational level of their parents.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Impact of exposure to television & electronic devices on attention in children. | baseline
  -Assessment of attention by Application of Gilliam 1995 for ADHD (numerical) (continous number) (>131 above high )-(130-131 high )-(111-130 above average )- (90-110 average)-(80-89 below average)-(70-79 low)-(<69 very low)
Exposure to television & electronic devices | baseline
  -Assess time of exposure by asking parents about Age of onset of screen exposure( in years)& duration of screen exposure( by hours).

SECONDARY OUTCOMES:
Impact of exposure to television& electronic devices on language development in children | baseline
  1-Assessment of receptive language in children
  * Application of Arabic language test (prepared by Nahla Abdelaziz Refaey 2004)(numerical)(continous number) (higher value 100 and lower value 0 , higher value is better outcome) 2-Assessment of expressive language development in children
  * Application of Arabic language test (prepared by Nahla Abdelaziz Refaey 2004)(numerical)(continous number) (higher value 100 and lower value 0 , higher value is better outcome) 3-Semantics score in language development in children
  * Application of Arabic language test (prepared by Nahla Abdelaziz Refaey 2004)(numerical)(continous number) (higher value 100 and lower value 0 , higher value is better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Sayed, professor, Study Chair — Assiut University; Abdallah Metwally, professor, Study Chair — Assiut University

REFERENCES:
- [Background] van den Heuvel M, Ma J, Borkhoff CM, Koroshegyi C, Dai DWH, Parkin PC, Maguire JL, Birken CS; TARGet Kids! Collaboration. Mobile Media Device Use is Associated with Expressive Language Delay in 18-Month-Old Children. J Dev Behav Pediatr. 2019 Feb/Mar;40(2):99-104. doi: 10.1097/DBP.0000000000000630. PMID 30753173
- [Background] Chonchaiya W, Pruksananonda C. Television viewing associates with delayed language development. Acta Paediatr. 2008 Jul;97(7):977-82. doi: 10.1111/j.1651-2227.2008.00831.x. Epub 2008 May 2. PMID 18460044
- [Background] Lin HP, Chen KL, Chou W, Yuan KS, Yen SY, Chen YS, Chow JC. Prolonged touch screen device usage is associated with emotional and behavioral problems, but not language delay, in toddlers. Infant Behav Dev. 2020 Feb;58:101424. doi: 10.1016/j.infbeh.2020.101424. Epub 2020 Feb 28. PMID 32120178
- [Background] Ruangdaraganon N, Chuthapisith J, Mo-suwan L, Kriweradechachai S, Udomsubpayakul U, Choprapawon C. Television viewing in Thai infants and toddlers: impacts to language development and parental perceptions. BMC Pediatr. 2009 May 22;9:34. doi: 10.1186/1471-2431-9-34. PMID 19460170
- [Background] Duch H, Fisher EM, Ensari I, Harrington A. Screen time use in children under 3 years old: a systematic review of correlates. Int J Behav Nutr Phys Act. 2013 Aug 23;10:102. doi: 10.1186/1479-5868-10-102. PMID 23967799
- [Background] Gentile DA, Oberg C, Sherwood NE, Story M, Walsh DA, Hogan M; American Academy of Pediatrics. Well-child visits in the video age: pediatricians and the American Academy of Pediatrics' guidelines for children's media use. Pediatrics. 2004 Nov;114(5):1235-41. doi: 10.1542/peds.2003-1121-L. PMID 15520101
- [Background] Domingues-Montanari S. Clinical and psychological effects of excessive screen time on children. J Paediatr Child Health. 2017 Apr;53(4):333-338. doi: 10.1111/jpc.13462. Epub 2017 Feb 6. PMID 28168778
- [Background] Harle B, Desmurget M. [Effects on children's cognitive development of chronic exposure to screens]. Arch Pediatr. 2012 Jul;19(7):772-6. doi: 10.1016/j.arcped.2012.04.003. Epub 2012 May 18. French. PMID 22609414
- [Background] Subrahmanyam K, Kraut RE, Greenfield PM, Gross EF. The impact of home computer use on children's activities and development. Future Child. 2000 Fall-Winter;10(2):123-44. PMID 11255703
- [Background] Christakis DA, Gilkerson J, Richards JA, Zimmerman FJ, Garrison MM, Xu D, Gray S, Yapanel U. Audible television and decreased adult words, infant vocalizations, and conversational turns: a population-based study. Arch Pediatr Adolesc Med. 2009 Jun;163(6):554-8. doi: 10.1001/archpediatrics.2009.61. PMID 19487612
- [Background] Tran P, Subrahmanyam K. Evidence-based guidelines for the informal use of computers by children to promote the development of academic, cognitive and social skills. Ergonomics. 2013;56(9):1349-62. doi: 10.1080/00140139.2013.820843. Epub 2013 Aug 7. PMID 23924039
- [Background] COUNCIL ON COMMUNICATIONS AND MEDIA. Media and Young Minds. Pediatrics. 2016 Nov;138(5):e20162591. doi: 10.1542/peds.2016-2591. PMID 27940793
- [Background] Radesky JS, Silverstein M, Zuckerman B, Christakis DA. Infant self-regulation and early childhood media exposure. Pediatrics. 2014 May;133(5):e1172-8. doi: 10.1542/peds.2013-2367. Epub 2014 Apr 14. PMID 24733868